CLINICAL TRIAL: NCT03193840
Title: Surgical Treatment of Old Acetabular Fracture With Posterior Wall Osteotomy
Brief Title: Posterior Wall Osteotomy for Old Acetabular Fracture
Acronym: osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRP1
Record Dates: First submitted 2017-06-11; First posted 2017-06-21 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Surgical Procedure, Unspecified
Keywords: old acetabular fracture; posterior wall osteotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- old acetabular fracture (Experimental): posterior wall osteotomy would be conducted for thr patient with displaced acetabular fracture without surgical treatment over three weeks.
  Interventions: Procedure: posterior wall osteotomy

INTERVENTIONS:
Procedure: posterior wall osteotomy — posterior wall osteotomy is conducted through Kocher-Langenbeck approach.

SUMMARY:
Posterior wall osteotomy would be conducted to manage the old acetabular fracture. The outcome was reviewed to assess the feasibility of the surgical procedure.

DETAILED DESCRIPTION:
More and more patients with old acetabular fracture were admitted in our institution during the past years. There is little literature especially depicts the therapeutic principle of the kind of damage. Posterior wall osteotomy would be conducted to eliminate the fragments or callus from the hip joint. Then, the deformed healing acetabulum could become mobile and the reduction may be achieved. However, the surgical procedure is technique demanding and some intraoperative risk may be accompanied.

Surgical time, blood loss, complication and fracture healing would be reviewed to assess the feasibility of the surgical procedure. The function outcome is evaluated with HHS score at the follow up.

ELIGIBILITY:
Inclusion Criteria:

* acetabular fracture
* no surgical procedure has been obtained over 3 weeks
* deformed healing
* receive posterior wall osteotomy
* completed more than one year follow-up

Exclusion Criteria:

* accompanied with other fracture
* pathological fracture
* reject the posterior wall osteotomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
frecture union time | 4 months
  the fracture line in the radiography

SECONDARY OUTCOMES:
complication | 1 month
  iatrogenic neurovascular injury

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Hou, Study Chair — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery
Locations (2):
- China (2):
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Zhiyong Hou, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No